CLINICAL TRIAL: NCT04748939
Title: Safety and Immunogenicity of a Recombinant Subunit Herpes Zoster Vaccine in Patients With Rheumatic Diseases Undergoing Immunosuppressive or Biologic/Targeted DMARD Therapies: a Double-blind Randomized Placebo-controlled Trial
Brief Title: Shingrix in Patients With Rheumatic Diseases: a Double-blind Placebo-controlled RCT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Dr, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NTWCShingrixstudy
Record Dates: First submitted 2021-02-07; First posted 2021-02-10 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Herpes Zoster
Keywords: vaccine; rheumatic diseases; immunosuppressive; immunogenicity; biologics; targeted DMARDs
MeSH Terms: conditions — Herpes Zoster; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: double-blind randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind for the identity of the drugs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vaccine (Active Comparator): Shingrix vaccine
  Interventions: Biological: recombinant subunit herpes zoster vaccine
- placebo (Placebo Comparator): normal saline injection (0.5mL)
  Interventions: Biological: recombinant subunit herpes zoster vaccine

INTERVENTIONS:
Biological: recombinant subunit herpes zoster vaccine — vaccine administration
  Other Names: Shingrix

SUMMARY:
A double-blind randomized controlled trial on the safety and immunogenicity of the recombinant subunit herpes zoster vaccine, Shingrix, in patients with rheumatic diseases undergoing immunosuppressive or biologic/targeted DMARD therapies

DETAILED DESCRIPTION:
A double-blind randomized controlled trial on the safety and immunogenicity of the recombinant subunit herpes zoster vaccine, Shingrix, in patients with rheumatic diseases undergoing immunosuppressive or biologic/targeted DMARD therapies.

Duration of study: 60 weeks

ELIGIBILITY:
Inclusion criteria for patients:

1. Patients with a diagnosis of rheumatic or immune-mediated diseases eg. SLE, RA, PSA, SpA, inflammatory myopathies, ANCA-related and large vessel vasculitides
2. Age ≥18 years
3. Stable or reducing doses of any the following immunosuppressive regimens within 4 weeks of study entry:

   1. Prednisolone ≥20mg/kg/day ± mycophenolate mofetil, azathioprine or the calcineurin inhibitors
   2. Cyclophosphamide (intravenous pulses or daily oral)
   3. B-cell depleting biological agents and their biosimilars eg. belimumab, anti-CD20 agents (next scheduled dose should be arranged to at least 12 weeks after study entry for rituximab or obinutuzumab)
   4. Anti-TNFα biological agents and their biosimilars eg. infliximab, etanercept, adalimumab, golimumab, certolizumab
   5. Anti-interleukin-6 biological agents eg. tocilizumab, sarilumab
   6. Other biological agents eg. abatacept, ustekinumab, secukinumab, ixekizumab
   7. The JAK inhibitors eg. tofacitinib, baricitinib, upadacitinib
4. Female patients with reproductive potential are allowed to participate in this study provided that they are willing to practice contraception for until at least 12 months after vaccination
5. Willing to comply with all study procedures

Exclusion criteria for patients:

1. Active infection, including upper respiratory tract infection
2. Active HZ infection
3. Active untreated tuberculosis
4. HIV infection
5. History of HZ or varicella vaccination in the past
6. History of allergy to any vaccines
7. Patients who are pregnant or plan to become pregnancy within one year of study entry
8. Lactating women
9. Patients who cannot give a written consent (mentally incapable or illiterate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
humoral immune response to Shingrix | week 12 (compared with baseline)
  proportion of patients with 4x fold increase in anti-gE antibody titer

SECONDARY OUTCOMES:
Humoral immune response | week 52
  proportion of patients with 4x fold increase in anti-gE antibody titer
adverse events | 7 days after injection
  solicited
adverse events | 4 weeks after injection
  unsolicited
flares of underlying diseases | week 26 and 60
  disease flares
herpes zoster infection | week 60
  herpes zoster infection
cell mediated response to vaccine | week 12 from baseline
  in 40 patients (20 from each arm); number of IFNγ-secreting CD4+ T cell colonies on ELISPOT assay

CONTACTS AND LOCATIONS:
Overall Officials: Chi Chiu Mok, Principal Investigator — Tuen Mun Hospital
Locations (1):
- Department of Medicine, Tuen Mun Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No